CLINICAL TRIAL: NCT03016806
Title: Umbilical Cord Blood Transplantation From Unrelated Donors
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Omar Aljitawi, Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Other Study IDs: UBMT 15029
Record Dates: First submitted 2016-12-26; First posted 2017-01-11 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Acute Leukemia; Immune Deficiency Disorder; Congenital Hematological Disorder; Metabolism Disorder; Aplastic Anemia; Myelodysplastic Syndromes; Chronic Leukemia; Lymphoma; Multiple Myeloma; Solid Tumor
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Metabolic Diseases; Anemia, Aplastic; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma | interventions — Cyclophosphamide; Mesna; Busulfan; fludarabine; Influenza Vaccines; Melphalan; Honey

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Full Intensity, TBI-based Conditioning: Full Intensity TBI-based Conditioning Total Body Irradiation 1200 cGy in fractions of 150 cGy days -8 or -7 to -4 Cyclophosphamide 60 mg/kg/day x 2 doses days -3 and -2 Mesna 60 mg/kg/day with 20% loading dose with first Cyclophosphamide followed by continuous infusion over 24 hours x 2 doses [to be completed 24 hours after final Cyclophosphamide dose] followed by Cord Blood Infusion Other names: TBI/Cy
  Interventions: Radiation: Total Body Irradiation 1200 cGy; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Cord Blood Infusion
- Full Intensity, Chemo-based Conditioning: Full Intensity, Chemotherapy Conditioning Busulfan days -7 to -4 Recipients <5 years - 1 mg/kg/dose x 16 doses every 6 hours Recipients >/= 5 years - 0.8 mg/kg/dose x 16 doses every 6 hours Cyclophosphamide 60 mg/kg/day x 2 doses days -3 and -2 Mesna 60 mg/kg/day with 20% loading dose with first Cyclophosphamide followed by continuous infusion over 24 hours x 2 doses [to be completed 24 hours after final Cyclophosphamide dose] followed by Cord Blood Infusion Other names: Bu/Cy
  Interventions: Drug: Cyclophosphamide; Drug: Mesna; Procedure: Cord Blood Infusion; Drug: Busulfan
- Reduced Intensity Chemotherapy: Reduced Intensity Chemotherapy Fludarabine 30 mg/m2/day x 5 doses days -6 to -2 Melphalan 140 mg/m2/day x 1 dose day -2 Cord Blood Infusion Other names: Flu/Mel
  Interventions: Procedure: Cord Blood Infusion; Drug: Fludarabine; Drug: Melphalan
- Non-Myeloablative Conditioning: Fludarabine 40 mg/m2/day x 5 doses days -6 to -2 Cyclophosphamide 50 mg/kg/day x 1 dose day -6 Mesna 50 mg/kg/day with 20% loading dose with Cyclophosphamide dose followed by continuous infusion over 24 hours x 1 dose [to be completed 24 hours after Cyclophosphamide dose] Total Body Irradiation 200 cGy in a single fraction day -1 Cord Blood Infusion Other names: Flu/Cy/TBI
  Interventions: Radiation: Total Body Irradiation 200 cGy; Drug: Cyclophosphamide; Drug: Mesna; Drug: Fludarabine

INTERVENTIONS:
Radiation: Total Body Irradiation 1200 cGy — Total Body Irradiation 1200 cGy in 8 fractions
  Other Names: TBI 1200 cGy
  Groups: Full Intensity, TBI-based Conditioning
Radiation: Total Body Irradiation 200 cGy — Total Body Irradiation 200 cGy in one fraction
  Other Names: TBI 200 cGy
  Groups: Non-Myeloablative Conditioning
Drug: Cyclophosphamide — 50 mg/kg or 60 mg/kg
  Other Names: Cy
  Groups: Full Intensity, Chemo-based Conditioning; Full Intensity, TBI-based Conditioning; Non-Myeloablative Conditioning
Drug: Mesna — 50 mg/kg or 60 mg/kg plus 10% loading dose
  Other Names: Pre-Mesna
  Groups: Full Intensity, Chemo-based Conditioning; Full Intensity, TBI-based Conditioning; Non-Myeloablative Conditioning
Procedure: Cord Blood Infusion — Intravenous infusion of cord blood stem cells
  Groups: Full Intensity, Chemo-based Conditioning; Full Intensity, TBI-based Conditioning; Reduced Intensity Chemotherapy
Drug: Busulfan — 0.8 mg/kg x 16 doses
  Other Names: Bu
  Groups: Full Intensity, Chemo-based Conditioning
Drug: Fludarabine — 30 mg/m2/day x 5 or 40 mg/m2/day x 5
  Other Names: Flu
  Groups: Non-Myeloablative Conditioning; Reduced Intensity Chemotherapy
Drug: Melphalan — 140 mg/m2
  Other Names: Mel
  Groups: Reduced Intensity Chemotherapy

SUMMARY:
This study is being done to determine how long it takes for the engraftment (recovery of blood cell counts) of umbilical cord stem cells and also how often engraftment of umbilical cord stem cells transplanted from an unrelated donor fails. Another purpose will be to document the rate of disease-free survival and the rate of relapse (a return of your disease or syndrome) as well as the incidence and severity of graft versus host disease (GvHD) following cord blood stem cell transplantation. GvHD is a complication of stem cell transplants in which white blood cells from the transplanted tissue (graft) attack the transplant recipient's body (host).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the kinetics of engraftment of umbilical cord blood (UCB) following transplantation into unrelated individuals.

II. Determine the incidence of non-engraftment and secondary graft failure when unrelated donor UCB cells are administered to patients receiving myeloablative, reduced intensity cytoreductive, or non-ablative conditioning regimens together with immunosuppressive therapy.

III. Determine the incidence and severity of graft-vs-host disease (GVHD) for patients receiving unrelated donor UCB grafts.

IV. Document the overall survival, disease-free-survival, and rates of relapse for UCB transplant recipients.

OUTLINE: This is an observational study.

Patients undergo a conditioning regimen per standard of care at the discretion of the treating provider, followed by a planned UCB transplantation on study. Patients also have their medical records reviewed for engraftment data on study.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate diagnosis: Patients must have a disease or syndrome amenable to therapy with hematopoietic stem cell transplantation. Diagnoses include, but are not limited to:
* Congenital and Other Non-malignant Disorders:
* Immunodeficiency disorders (e.g. Severe Combined Immunodeficiency, Wiskott-Aldrich Syndrome)
* Congenital hematopoietic stem cell defects (e.g. Chediak-Higashi Syndrome, Congenital Osteopetrosis, Osteogenesis Imperfecta)
* Metabolic disorders (e.g. Hurler's Syndrome)
* Severe aplastic anemia
* High-Risk Leukemia:
* Acute Myelogenous Leukemia
* Refractory to standard induction therapy (more than 1 cycle required to achieve remission)

  * Recurrent (in CR ≥ 2)
  * Treatment-related AML or MDS
  * Evolved from myelodysplastic syndrome
  * Presence of FLT3 abnormalities
  * FAB M6 or M7
  * Adverse cytogenetics
  * Myelodysplastic Syndrome
  * Acute Lymphoblastic Leukemia including T lymphoblastic leukemia:
  * Refractory to standard induction therapy (time to CR >4 weeks)
  * Recurrent (in CR ≥ 2)
  * WBC count >30,000/mcL at diagnosis
  * Age >30 at diagnosis
* Adverse cytogenetics, such as t(9:22), t(1:19), t(4:11), and other MLL rearrangements.
* Chronic Myelogenous Leukemia in accelerated phase or blast crisis
* Biphenotypic or undifferentiated leukemia
* Burkitt's leukemia or lymphoma
* Lymphoma:
* Large cell, Mantle cell, Hodgkin lymphoma refractory or recurrent, chemo-sensitive, and ineligible for an autologous stem cell transplant or previously treated with autologous SCT
* Marginal zone or follicular lymphoma that is progressive after at least two prior therapies
* Multiple Myeloma, recurrent following high-dose therapy and autologous SCT or ineligible for an autologous HSCT
* Solid tumors, with efficacy of allogeneic HSCT demonstrated for the specific disease and disease status
* Adequate organ function:
* Cardiac - LVEF >45%, or shortening fraction >25%, Absence of congestive heart failure or conduction disturbances with high risk for sudden death
* Pulmonary - DLCO (corrected for hemoglobin), FEV1 and FVC ≥ 50% predicted;
* Renal - serum Cr < 1.5 times the upper limit of normal for age or GFR ≥ 50 ml/min/1.73m2
* Hepatic - total bilirubin level < 2 times the upper limit of normal (except for patients with Gilbert's syndrome or hemolysis); if the primary disease process is causal, this criterion will be reconsidered. ALT, AST, and Alkaline phosphatase ≤ 5 times upper limit of normal.
* Performance Status Karnofsky or Lansky score ≥ 70%.
* Informed Consent must be obtained prior to initiating conditioning therapy.
* Receipt of viable cord blood product(s), single or dual, must be confirmed with the stem cell processing laboratory prior to initiating conditioning therapy.

Exclusion Criteria:

* Availability of 10/10 or 9/10 HLA-matched related or unrelated donor within a reasonable timeframe dictated by the clinical urgency of the transplant
* Autologous HSCT < 6 months prior to proposed UCB transplant
* Pregnant or breast feeding
* Current uncontrolled infection
* Evidence of HIV infection or positive HIV serology

Ages: 2 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Engraftment of ANC and Platelets | 42 days following the infusion of stem cells for ANC [If engraftment of ANC does not occur within 42 days, a subsequent transplant will be performed if a donor is available.]
  The date of engraftment of ANC is the first of 3 consecutive days of ANC of 500 or higher based on daily CBC and Differential Counts. The date of engraftment of platelets is the first of three consecutive days of platelet counts of 20,000 or higher in the absence of platelet transfusions for a t least 7 days prior.

SECONDARY OUTCOMES:
Rate of non-engraftment and of secondary graft failure | At 30 days, 100 days, 6 months and yearly from the date of transplant until the date of documented graft failure or the subject's death up to 120 months.
  The percentage of patients who fail to initially engraft ANC will be tabulated as well as the percentage of patients who have primary engraftment of ANC but whose graft fails as evidenced by pancytopenia, failure of bone marrow function and loss of donor chimerism following initial engraftment of ANC.
Incidence of acute graft-versus-host disease | At 30 days and 100 days after transplant from the date of transplant until the date of documented acute GvHD.
  Routine physical exams, liver function tests, and clinical history of diarrhea and upper GI symptoms will be used to assess the presence of, the maximum severity of and the date of onset of Acute GvHD based on the criteria published by Przepioka et al., Bone Marrow Transplant 1995; 15(6):825-8 as used by the Center for International Blood & Marrow Transplant Research. The percentage of patients developing symptoms of acute graft-versus-host disease will be tabulated.
Incidence of chronic graft-versus-host disease | At 100 days, 6 months and yearly after transplant from the date of transplant until the date of documented graft failure or the subject's death up to 120 months.
  Assess the presence of and the maximum severity of and the date of onset of chronic GvHD based on Sullivan KM, Blood 1981;57-267 as used by the Cneter for International Blood & Marrow Transplant Research.
Disease-free survival | At 30 days, 100 days, 6 months and yearly after transplant from the date of transplant until the date of documented graft failure or the subject's death up to 120 months.
  Document and update the length of time a subject survives without recurrence of the disease for which they were transplanted at 30 days, 100 days, 6 months and yearly following the infusion of cord blood stem cells for as long as the subjects survive and remain disease-free.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — Professor - Department of Medicine, Hematology/Oncology (SMD)
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No